CLINICAL TRIAL: NCT03584958
Title: Comparing Refractive and Visual Outcomes of Minimally Invasive and Traditional Glaucoma Surgeries
Brief Title: Comparing Refractive and Visual Outcomes of MIGS and Traditional Surgeries
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Wills Eye (Other)
Collaborators: Allergan (Industry); The American Society of Cataract and Refractive Surgery Foundation (Other)
Responsible Party: Principal Investigator, Daniel Lee, MD, Principal Investigator, Wills Eye
Other Study IDs: 18-689E
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: glaucoma surgery; MIGS, minimally invasive glaucoma surgery; refractive outcomes; visual outcomes
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Ab interno goniotomy surgery: Gonioscopy-assisted transluminal trabeculotomy (GATT) surgery to decrease intraocular pressure.
- Gelatin stent surgery: Subconjunctival stent (Xen) surgery to decrease intraocular pressure.
- Suprachoroid stent and cataract surgery: Suprachoroidal stent (Cypass) to decrease intraocular pressure in combination with cataract surgery.
- Trabeculectomy surgery: Glaucoma filtering surgery to decrease intraocular pressure.
- Cataract surgery: Cataract surgery with no glaucoma procedure.

SUMMARY:
The primary goal of this study is to evaluate refractive and visual outcomes in glaucoma patients who will be having either traditional glaucoma surgery or minimally invasive glaucoma surgery, also known as MIGS.

DETAILED DESCRIPTION:
There is an increasing number of surgical options to lower intraocular pressure (IOP) in patients with glaucoma and ocular hypertension performed with or without concurrent cataract surgery. Today, patients undergoing glaucoma surgery have increasingly higher expectations for their postoperative visual outcomes. Therefore, it is important to understand the influence of various glaucoma surgical procedures on refractive outcomes. This information would aid in patient and surgical procedure selection, pre-operative counseling to set appropriate expectations and may help surgeons adjust their plans and techniques to improve visual outcomes.

The advent of minimally invasive glaucoma surgery (MIGS) procedures further highlights the importance of studying refractive outcomes as many of these surgeries are being performed earlier in the glaucoma severity spectrum where central visual potential is still preserved. Furthermore, this class of surgeries is often performed in combination with cataract surgery.

There remains a lack of data regarding refractive outcomes in patients who have had phaco-iStent, phaco-Cypass, as well as goniotomy (Kahook dual blade (KDB) gonioscopy assisted transluminal trabeculotomy), and Xen gel stent implantation with or without cataract surgery. This information would help during pre-operative patient discussions and lens selection in the context of a combined procedure.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of glaucoma or ocular hypertension in the study eye(s) and are consented to receive any of the following procedures:

* Ab interno goniotomy surgery: Gonioscopy-assisted transluminal trabeculotomy (GATT) surgery to decrease intraocular pressure.
* Gelatin stent surgery: Subconjunctival stent (Xen) surgery to decrease intraocular pressure.
* Suprachoroidal stent and cataract surgery: Suprachoroidal stent (Cypass) to decrease intraocular pressure in combination with cataract surgery.
* Trabeculectomy surgery: Glaucoma filtering surgery to decrease intraocular pressure.
* Cataract surgery: Cataract surgery with no glaucoma procedure.

Exclusion Criteria:

Patients with previous corneal ectasia or history of refractive procedures; patients who cannot fixate well due to poor vision (worse than 20/200)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Wills Eye Hospital Glaucoma Service who are in need of glaucoma and/or cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Biometry prediction accuracy | Baseline, Post-op Month 1, Post-op Month 3
  Difference between the target refraction and the spherical equivalent of the final refraction following surgery.

SECONDARY OUTCOMES:
Post-operative corneal curvature | Baseline, Post-op Month 1, Post-op Month 3
  Variation in corneal curvature (astigmatism) following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lee, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No